CLINICAL TRIAL: NCT05951725
Title: A Randomized, Blinded, Positive Vaccine-controlled Phase III Clinical Trial to Evaluate the Safety and Immunogenicity of DTcP in Infants and Children at 2 and 3 Months of Age
Brief Title: A Clinical Trial of Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed(DTcP)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CS-CTP-DTcP-Ⅲ
Record Dates: First submitted 2023-07-02; First posted 2023-07-19 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Diphtheria, Tetanus and Acellular Pertussis
Keywords: Vaccine; Three Components; Immunogenicity; Safety
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Tetanus Toxoid; Vaccines, Combined; diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental vaccine group A，3 months old (Experimental): 4 doses of DTcP vaccine (0.5 ml) on Day 0 and Month 1,2,15~21
  Interventions: Biological: Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed (DTcP)
- Control vaccine group B，3 months old (Active Comparator): 4 doses of DTaP vaccine (0.5 ml) on Day 0 and Month 1,2,15~21
  Interventions: Biological: Diphtheria，Tetanus and Acellular Pertussis Combined Vaccine，DTaP
- Control vaccine group C，3 months old (Active Comparator): 4 doses of DTaP-IPV-Hib vaccine (0.5 ml) on Day 0 and Month 1,2,15~21
  Interventions: Biological: Diphtheria,tetanus,pertussis(acellular,component),Inactivated polio vaccine(adsorbed）and Haemophilus influenzae type b conjugate vaccine,adsorbed,DTaP-IPV-Hib
- Experimental vaccine group D，2 months old (Experimental): 4 doses of DTcP vaccine (0.5 ml) on Day 0 and Month 1,2,16~22
  Interventions: Biological: DTcP
- Control vaccine group E，2 months old (Active Comparator): 4 doses of DTaP-IPV-Hib vaccine (0.5 ml) on Day 0 and Month 1,2,16~22
  Interventions: Biological: DTaP-IPV-Hib
- Experimental vaccine group F，2 months old (Experimental): 4 doses of DTcP vaccine (0.5 ml) on Day 0 and Month 2,4,16~22
  Interventions: Biological: DTcP

INTERVENTIONS:
Biological: Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed (DTcP) — Three doses of basic immunization were completed at 3, 4 and 5 months of age, and one dose of booster immunization was completed at 18 to 24 months of age.
  Arms: Experimental vaccine group A，3 months old
Biological: Diphtheria，Tetanus and Acellular Pertussis Combined Vaccine，DTaP — Three doses of basic immunization were completed at 3, 4 and 5 months of age, and one dose of booster immunization was completed at 18 to 24 months of age.
  Arms: Control vaccine group B，3 months old
Biological: Diphtheria,tetanus,pertussis(acellular,component),Inactivated polio vaccine(adsorbed）and Haemophilus influenzae type b conjugate vaccine,adsorbed,DTaP-IPV-Hib — Three doses of basic immunization were completed at 3, 4 and 5 months of age, and one dose of booster immunization was completed at 18 to 24 months of age.
  Arms: Control vaccine group C，3 months old
Biological: DTcP — Three doses of basic immunization were completed at 2, 3 and 4 months of age, and one dose of booster immunization was completed at 18 to 24 months of age.
  Arms: Experimental vaccine group D，2 months old
Biological: DTaP-IPV-Hib — Three doses of basic immunization were completed at 2, 3 and 4 months of age, and one dose of booster immunization was completed at 18 to 24 months of age.
  Arms: Control vaccine group E，2 months old
Biological: DTcP — Three doses of basic immunization were completed at 2, 4 and 6 months of age, and one dose of booster immunization was completed at 18 to 24 months of age.
  Arms: Experimental vaccine group F，2 months old

SUMMARY:
The combined pertussis, diphtheria and tetanus vaccine, the first vaccine to be included in the Expanded Programme of Immunization(EPI) of World Health Organization(WHO), has played an important role in the prevention and control of these three infectious diseases. The (diphtheria，tetanus and acellular pertussis combined vaccine，DTaP) vaccine was successfully developed in China in 1993, and its safety and serological effects were confirmed by the observation of human safety, with mild vaccination reactions and good immunization effects.The (Diphtheria-tetanus-component acellular pertussis vaccine, DTcP) vaccine is suitable for immunization against pertussis, diphtheria and tetanus infections in people between 2 and 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* 2 months of age (60~89 days), 3 months of age (90~119 days), willing to provide identification documents
* The legal guardian or delegate has given informed consent, voluntarily signed the informed consent form, and can comply with the requirements of the clinical study protocol

Exclusion Criteria:

* Infants 2 months of age who have received a vaccine containing the components of diphtheria, IPV, Hib, or 13-valent pneumococcal polysaccharide conjugate vaccine
* Infants 3 months of age who have received vaccines containing diphtheria, Hib, or 13-valent pneumococcal polysaccharide conjugate vaccine or group A, group C meningococcal conjugate vaccine
* 3-month-old infant vaccinated with IPV
* Premature birth (delivery before the 37th week of gestation), low birth weight (birth weight <2500g) for 2-month-old (60-89 days) and 3-month-old (90-119 days) infants
* History of abnormal labor, asphyxia, and neurological damage
* Those who have suffered from pertussis, diphtheria or tetanus
* Individuals who have had household contact with individuals with confirmed pertussis, diphtheria, or tetanus disease in the past 30 days
* History of allergy to vaccines or vaccine components, severe side effects to vaccines such as allergy, urticaria, respiratory distress, angioneurotic edema
* Those with a history of epilepsy, convulsions, convulsions, cerebral palsy, or a history of mental illness or family history; or other progressive neurological disorders
* Have been diagnosed with a congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), juvenile rheumatoid arthritis (JRA), or other autoimmune disease
* Any condition resulting in absence of spleen, defective spleen function
* Known or suspected acute disease or serious chronic disease (including: serious respiratory disease, serious cardiovascular disease, liver and kidney disease, serious skin disease, malignant tumor, etc.); or in the acute phase of chronic disease
* Physician-diagnosed coagulation abnormalities (e.g., clotting factor deficiency, coagulopathy, platelet abnormalities) or significant bruising or clotting disorders
* Have had immunosuppressive or modifying agents, cytotoxic continuous treatment for more than 10 days in the past 6 months (except inhaled and topical steroids)
* Received blood products (except hepatitis B immunoglobulin) within 3 months prior to receiving the experimental vaccine
* Received another investigational drug or investigational vaccine within 1 month prior to receiving the experimental vaccine
* Plan to participate or are participating in any other drug clinical studies
* Received a live attenuated vaccine within 14 days prior to receiving the experimental vaccine, or received another vaccine within 7 days
* Those with fever before vaccination, axillary body temperature >37.0°C
* Any other factors that, in the judgment of the investigator, make participation in the clinical trial inappropriate
* 1-20 articles for the first dose exclusion criteria
* Those who had a severe allergic reaction after the previous dose of vaccine
* Persons with serious adverse reactions causally related to the previous dose of vaccination
* Newly discovered or newly occurred after the first vaccination that do not meet the first dose inclusion criteria or meet the first dose exclusion criteria will be determined by the investigator whether to continue to participate in the study
* Other reasons for exclusion as perceived by the researcher
* 22-25 for the 2nd, 3rd, 4th agent exclusion criteria

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2520 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Serum anti-Pertussis Toxoid(PT), Filamentous hemagglutmin(FHA), Pertactin(PRN), DT(Diphtheria Toxoid), TT(Tetanus Toxoid) antibody positive conversion rate,GMC 30 days after completion of basal immunization in subjects in the 3-month-old group | 30 days after completion of basal immunization
Serum anti-PT, FHA, PRN, DT, TT antibody positive conversion rate, Geometric Mean Concentration(GMC) 30 days after completion of basal immunization in subjects in the 2-month-old group | 30 days after completion of basal immunization
Incidence of adverse reactions within 0-30 days after each dose of vaccination in subjects in the 3-month-old group | Within 0-30 days after each dose of vaccination
Incidence of adverse reactions within 0-30 days after each dose of vaccination in subjects in the 2-month-old group | Within 0-30 days after each dose of vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Changge Center for Disease Control and Prevention, Xuchang, Henan, China